CLINICAL TRIAL: NCT00838292
Title: Randomized Controlled Evaluation of the Impact of Food Supplements on Malnourished HIV-Infected Adult ART Clients and Malnourished, HIV-Infected Pre-ART Adults in Kenya
Brief Title: Study of Impacts of Food Supplementation on Malnourished HIV-Infected Adults in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academy for Educational Development (Industry)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Robert Mwadime and Tony Castleman, Academy for Educational Development, FANTA Project
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AED 1
Record Dates: First submitted 2009-02-03; First posted 2009-02-06 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-02

CONDITIONS: HIV; Malnutrition; HIV Infections
Keywords: food supplementation; HIV; malnutrition
MeSH Terms: conditions — Malnutrition; HIV Infections | interventions — Pharmaceutical Preparations; Whey

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ART: food (Active Comparator): ART + food supplementation + nutrition counseling
  Interventions: Dietary Supplement: fortified blended flour - Insta Foundation Plus (with whey protein concentrate); Other: nutrition counseling
- ART: no food (Active Comparator): ART + nutrition counseling
  Interventions: Other: nutrition counseling
- pre-ART: food (Active Comparator): no ART (cotrimoxazole provided) + food supplementation + nutrition counseling
  Interventions: Dietary Supplement: fortified blended flour - Insta Foundation Plus (with whey protein concentrate); Other: nutrition counseling
- pre-ART: no food (Active Comparator): no ART (cotrimoxazole provided) + nutrition counseling
  Interventions: Other: nutrition counseling

INTERVENTIONS:
Dietary Supplement: fortified blended flour - Insta Foundation Plus (with whey protein concentrate) — 300 grams/day for 6 months
  Other Names: Insta Products Ltd. Foundation Plus product with whey protein concentrate.
  Arms: ART: food; pre-ART: food
Other: nutrition counseling

SUMMARY:
The purpose of the study is to test whether food supplementation of malnourished HIV-infected adults (both pre-ART and ART) in resource constrained settings improves their nutritional status, clinical status, effectiveness of treatment, quality of life, functioning, and survival.

DETAILED DESCRIPTION:
Malnutrition remains a significant problem among HIV-infected populations, even among those with access to ART. In patients with HIV infection, poor nutritional status is associated with significant reduction in survival rates, accelerated disease progression, diminished response to therapies including ART, increased susceptibility to opportunistic infections, and reduced work capacity and quality of life. However, there is not evidence whether delay or reversal of weight loss improves life expectancy, nor is there evidence about the specific benefits food supplementation has on people with HIV infection. As antiretroviral therapy (ART) services continue to scale up in sub-Saharan Africa, there is a critical need for information about the impacts of appropriate food supplementation on the effectiveness of ART, on the health status of clients, and on the progression of the disease.

Malnourished adult ART and pre-ART clients at six clinical sites in Kenya are randomly allocated either to a group that receives nutrition counseling only or a group that receives nutrition counseling and supplementary feeding for six months. All patients continue to receive medical treatment (ART and other medicine) according to their condition. Baseline measures of socioeconomic and demographic status are collected. Measures of both nutritional and non-nutritional clinical outcomes are collected at baseline, 3, 6, 9, and 12 months. Clients beginning ART are treated as one arm and randomized between food and non-food, and clients not yet eligible for ART (pre-ART) are treated as a second arm and randomized between food and non-food. Within each arm, outcomes of subjects receiving supplemental food will be compared with outcomes of those who are not.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* BMI < 18.5
* Resident of area for past 6 months

Exclusion Criteria:

* Pregnant or lactating (child < 6 months)
* BMI > 18.5, BMI < 14
* Already receiving other food supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Body Mass Index | monthly

SECONDARY OUTCOMES:
CD4 counts | every three months (quarterly)
Quality of Life | monthly
drug adherence | monthly

CONTACTS AND LOCATIONS:
Overall Officials: James Muttunga, Ph.D., Principal Investigator — Kenya Medical Research Institute; Robert Mwadime, Ph.D., Principal Investigator — Academy for Educational Development, FANTA Project
Locations (6):
- Kenya (6):
  - Maragwa District Hospital, Maragwa
  - Mathere North Hospital, Nairobi
  - Mbagathi District Hospital, Nairobi
  - Riruta City Council Hospital, Nairobi
  - Naivasha District Hospital, Naivasha
  - Nyeri Provincial Hospital, Nyeri